CLINICAL TRIAL: NCT00068432
Title: A Phase II Trial of Gemcitabine and Celecoxib as First-Line Treatment for Patients With Advanced Metastatic Pancreatic Cancer
Brief Title: Gemcitabine and Celecoxib in Treating Patients With Metastatic Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2003-0288; P30CA016672 (NIH); MDA-2003-0288 (Other: UT MD Anderson Cancer Center); NCI-6167; CDR0000322827 (Registry Identifier: NCI PDQ)
Record Dates: First submitted 2003-09-10; First posted 2003-09-11 (Estimated); Last update posted 2018-10-31 (Actual); Status verified 2018-10

CONDITIONS: Pancreatic Cancer
Keywords: recurrent pancreatic cancer; stage IV pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Celecoxib; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Gemcitabine + Celecoxib (Experimental): Oral celecoxib twice daily on days 1-28. Gemcitabine by vein (IV) over 65 minutes on days 1, 8 and 15. Courses repeat every 4 weeks.
  Interventions: Drug: Celecoxib; Drug: Gemcitabine Hydrochloride

INTERVENTIONS:
Drug: Celecoxib — Oral celecoxib twice daily on days 1-28. Courses repeat every 4 weeks.
  Other Names: Celebrex
Drug: Gemcitabine Hydrochloride — Receive gemcitabine by vein (IV) over 65 minutes on days 1, 8 and 15. Courses repeat every 4 weeks.
  Other Names: Gemcitabine; Gemzar

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as gemcitabine, use different ways to stop tumor cells from dividing so they stop growing or die. Celecoxib may stop the growth of pancreatic cancer by stopping blood flow to the tumor and blocking the enzymes necessary for tumor cell growth. Combining gemcitabine with celecoxib may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving gemcitabine together with celecoxib works in treating patients with metastatic pancreatic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the overall survival at 6 months in patients with metastatic pancreatic cancer treated with gemcitabine and celecoxib.
* Determine the objective tumor response, progression-free survival, and median survival of patients treated with this regimen.
* Determine the safety and toxicity of this regimen in these patients.

OUTLINE: This is a nonrandomized, open-label, multicenter study.

Patients receive gemcitabine IV over 65 minutes on days 1, 8, and 15 and oral celecoxib twice daily on days 1-28. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.

Patients are followed monthly for 6 months from study entry and then every 3 months thereafter.

PROJECTED ACCRUAL: A total of 40 patients will be accrued for this study within 8 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed metastatic pancreatic cancer
* Radiographic evidence of disease
* No known brain metastases

PATIENT CHARACTERISTICS:

Age

* Any age

Performance status

* ECOG 0-2 OR
* Karnofsky 60-100%

Life expectancy

* Not specified

Hematopoietic

* WBC at least 3,000/mm^3
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic

* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* AST/ALT no greater than 2.5 times ULN

Renal

* Creatinine normal OR
* Creatinine clearance at least 60 mL/min

Cardiovascular

* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia

Gastrointestinal

* No history of peptic ulcer disease
* No gastrointestinal bleeding within the past 3 months

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No prior allergic reactions to compounds of similar chemical or biological composition to study drugs or to sulfonamides
* No prior allergic reaction, asthma, or urticaria after taking aspirin or NSAIDs
* No ongoing or active infection
* No other uncontrolled illness
* No psychiatric illness or social situation that would preclude study compliance
* No other malignancy within the past 5 years except basal cell skin cancer or carcinoma in situ of the cervix

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* No prior chemotherapy for metastatic pancreatic cancer
* More than 6 months since prior neoadjuvant or adjuvant chemoradiotherapy (including gemcitabine) for pancreatic cancer

Endocrine therapy

* Not specified

Radiotherapy

* See Chemotherapy
* More than 6 months since prior radiotherapy

Surgery

* Not specified

Other

* More than 30 days since prior investigational agents
* No other concurrent investigational or commercial agents or therapies for the malignancy
* No other concurrent nonsteroidal anti-inflammatory drugs (NSAIDs)
* No other concurrent cyclo-oxygenase-2 (COX-2) inhibitors (e.g., rofecoxib)
* Concurrent acetaminophen-containing medications or low-dose aspirin (up to 325 mg/day) for cardiac prophylaxis allowed

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2003-12; Primary Completion 2005-07 (Actual); Study Completion 2005-07 (Actual)

PRIMARY OUTCOMES:
Overall Survival at 6 months | 6 Months

SECONDARY OUTCOMES:
Overall response rate | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Henry Q. Xiong, MD, PhD, Principal Investigator — M.D. Anderson Cancer Center
Locations (11):
- United States (11):
  - Hembree Mercy Cancer Center at St. Edward Mercy Medical Center, Fort Smith, Arkansas
  - M.D. Anderson Cancer Center - Orlando, Orlando, Florida
  - CCOP - Atlanta Regional, Atlanta, Georgia
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - CCOP - Wichita, Wichita, Kansas
  - CCOP - Kansas City, Kansas City, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - CCOP - Dayton, Dayton, Ohio
  - CCOP - Columbia River Oncology Program, Portland, Oregon
  - M.D. Anderson Cancer Center at University of Texas, Houston, Texas
  - All Saints Cancer Center at All Saints Healthcare, Racine, Wisconsin

REFERENCES:
- See also: UT MD Anderson Cancer Center Website — http://www.mdanderson.org